CLINICAL TRIAL: NCT02042586
Title: Evaluation of Locomotor Activity Before and After Total Hip Replacement in Patients With Hip Osteoarthritis. Use of Ganglion and Neural Network Techniques to Identify Objective Criteria for the Success of Arthroplasty
Brief Title: Evaluation of Locomotor Activity Before and After Total Hip Replacement in Patients With Hip Osteoarthritis.
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: TROUILLOUD AOI 2007
Record Dates: First submitted 2014-01-17; First posted 2014-01-23 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Hip Osteoarthritis; Indication for Total Hip Replacement
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Patients
  Interventions: Other: Analysis of movement before total hip replacement; Other: Analysis of movement after total hip replacement
- Controls
  Interventions: Other: Analysis of movement before total hip replacement

INTERVENTIONS:
Other: Analysis of movement before total hip replacement
Other: Analysis of movement after total hip replacement
  Groups: Patients

SUMMARY:
The investigators believe that the application of non-linear methods of analysis using the ganglion and neural network technique will make it possible to analyse all of the complex data obtained in patients with hip osteoarthritis before and then after total hip replacement, and should allow us to identify a combination of objective variables to classify the surgery as " successful " or " unsuccessful ".

To this end, the study will take place as follows:

Step 1: Screening, and inclusion. Step 2: Evaluation of the hip osteoarthritis and analysis of locomotor activity Step 3: Total hip replacement Step 4: Clinical evaluation of locomotor activity carried out between 6 months and 1 year after the THR Step 5: Data analysis

ELIGIBILITY:
Inclusion Criteria:

Control group:

* Subjects who have provided written informed consent
* Subjects covered by the national health insurance scheme
* Men or women aged between 25 and 85 years
* able to understand simple instructions and packaging instructions and able to give informed consent

Patients group:

* Patients who have provided written informed consent
* Patients covered by the national health insurance scheme
* Men or women aged between 25 and 85 years
* able to understand simple instructions and packaging instructions and to give their informed consent
* Suffering from hip osteoarthritis defined according to ACR criteria
* Most recent radiography examination less than 6 months earlier
* Radiological stage II, III or IV hip osteoarthritis according to the Kellgren and Lawrence classification
* Presenting with an indication for total hip replacement, according to the surgeon's usual criteria

Exclusion Criteria:

Control group:

* Hip osteoarthritis or other arthrosis in the lower limbs
* Pregnant or breast-feeding women
* Disorders that may interfere with gait analysis
* Disorder that may be destabilized by gait analysis
* Neurological disease and/or motor neuron disease

Patients group:

* Contra-indication for total hip replacement
* Repeat surgery for total hip replacement
* Impossibility to use a standard implant
* Pregnant or breast-feeding women
* Inflammatory flare of the hip osteoarthritis
* Disorder that may interfere with gait analysis
* Disorder that may be destabilized by gait analysis
* Rapidly destructive hip osteoarthritis
* Neurological disease and/or motor neuron disease
* Hip dysplasia requiring THR to be completed using a graft

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: hip osteoarthritis indication for total hip replacement
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2010-01-07 (Actual); Primary Completion 2014-12-11 (Actual)

PRIMARY OUTCOMES:
Degree of patient statisfaction | Before and between 6 months and 1 year after total hip replacement

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de DIJON, Dijon, France

REFERENCES:
- [Derived] Riglet L, Bourredjem A, Laroche D, Benguella L, Binquet C, Maillefert JF, Ornetti P, Gueugnon M. Hip disability and Osteoarthritis Outcome Score trajectories and prognostic factors for functional decline: A 3-year follow-up study. Ann Phys Rehabil Med. 2025 Feb;68(1):101893. doi: 10.1016/j.rehab.2024.101893. Epub 2024 Dec 9. PMID 39657458
- [Derived] Moissenet F, Naaim A, Ornetti P, Bourredjem A, Binquet C, Morisset C, Gouteron A, Maillefert JF, Laroche D. Is the Pelvis-Thorax Coordination a Valuable Outcome Instrument to Assess Patients With Hip Osteoarthritis? Front Bioeng Biotechnol. 2020 Jan 23;7:457. doi: 10.3389/fbioe.2019.00457. eCollection 2019. PMID 32039174